CLINICAL TRIAL: NCT07030998
Title: WEARABLES: Wearable Technology and Machine Learning for Early Detection and Risk Assessment of Unacceptable Toxicities in a Paediatric Oncology Cohort
Brief Title: Wearable Technology and Machine Learning for Early Detection and Risk Assessment of Unacceptable Toxicities in a Paediatric Oncology Cohort
Acronym: WEARABLES
Status: Recruiting | Type: Observational
Sponsor: Murdoch Childrens Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 111206
Record Dates: First submitted 2025-05-15; First posted 2025-06-22 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Cancer; Infection; Digital Health; Wearable Devices
Keywords: Cancer; Paediatric; Infection; Treatment Toxicity; Wearable Device
MeSH Terms: conditions — Neoplasms; Infections | interventions — Wearable Electronic Devices

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Wearable Device — Wearable device to collect the following health metrics directly from participants for the duration of the study (4 weeks). Health metrics are collected every 15 minutes, except for the ECG which will be collected once per week.
  Data points:
  * ECG data (Once per week)
  * Exercise time
  * Body Temperature
  * Heart Rate
  * Irregular Heart Rhythm
  * Blood Oxygen Saturation
  * Respiratory Rate

SUMMARY:
Data collection study to establish a predictive model of infection observed during childhood cancer therapy using data captured by wearable technology.

DETAILED DESCRIPTION:
Rationale: Development in treatment for childhood cancers has improved remarkably with the 5-year survival rate now exceeding 80% in developed countries. However, these treatments are not without their adverse effects. The international Childhood Cancer Survivor study revealed that 62.3% of survivors had at least one chronic health condition and 27.5% had a severe or life-threatening condition as a direct result of their cancer treatment (DOI: 10.1056/NEJMsa060185). One of the adverse events experienced by 90% of children treated for cancer is infection. Septic shock, the most severe of infection outcomes, is characterized by life-threatening organ dysfunction, is the most and carriers a mortality rate of 41 to 46% (DOI: 10.1016/j.jped.2023.01.001). Beyond mortality, delayed first antibiotic administration (> 1 hour from fever onset >38 degrees) is associated with intensive care admissions, prolonged hospital stays, and adverse outcomes. Fluctuations in physiology can precede fever onset by 72 hours in patients with infection. This may provide a window for early detection of infection via wearable technology. The WEARABLES study will combine wearable technology with machine learning to develop an infection prediction model to allow earlier detection and reduce the suffering of children with cancer.

Trial Design: This is a non-interventional silent pilot trial to establish a predictive model for infection observed during childhood cancer therapy using data passively captured via wearables.

The study will be conducted in patients (5-18 years) with a new cancer diagnosis, currently receiving treatment at The Royal Children's Hospital, and have access to an iPhone (either themselves as an adolescent and young adult or via their parents/guardian). Once consented the wearable device will be paired to the patients or parent/guardians phone, and the WEARABLES app will be downloaded onto the phone. Once the device has been set up correctly, the wearable device will collect a range of vital signs for the duration of the study (4 weeks), and a weekly survey will be sent to check for symptoms and/or hospital admissions for infection. At the end of the 4 weeks, participants will receive a final survey to evaluate the feasibility of using a wearable device for toxicity detection. No further involvement will be asked of participants for this pilot trial. All data collected will be utilized to develop a machine learning model for sepsis/infection before being prospectively validated in a second trial.

ELIGIBILITY:
Inclusion Criteria:

* Paediatric, adolescent or young adult diagnosis of cancer AND receiving therapy placing them at risk of infection
* Receiving cancer treatment at The Royal Children's Hospital
* Patients aged 5-18 years at time of the eligibility screening
* If aged < 16 years, parent or guardian able to provide consent
* iPhone 8 or later (iOS must be up to date/updated at time of enrolment)
* At least 10MB of iPhone storage for WEARABLES app and data collection.
* Willing and able to wear a wearable device for a period of 4 weeks (during waking hours).
* Consent to data being shared to the WEARABLES app (owned by the research team).

Exclusion Criteria:

* <5 years of age.
* <16 years of age without guardian or parent consent.
* Aged 16-18 and unable to provide consent.
* Participant did not consent to wearing Apple Watch for a period of 4 weeks.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients aged 5-18 years currently receiving treatment for cancer at The Royal Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Changes in cardiac electrical activity patterns on Electrocardiogram (ECG) | Baseline (Day 1), Day 8, Day 15, Day 22, Day 29
  ECG data will be collected once per week over a 4-week period for each participant to identify changes in cardiac electrical activity that may be associated with early infection. These data will be used as input features for a machine learning model aimed at predicting infection risk in children receiving cancer treatment.
Changes in physical activity | Baseline (Day 1) and every 15 minutes until Study completion at Day 29
  Exercise data will be collected every 15 minutes over a 4-week period for each participant to identify changes that may correlate with early signs of infection. These data points will be used as input features for a machine learning model aimed at predicting infection risk in children receiving cancer treatment.
Changes in heart rate | Baseline (Day 1) and every 15 minutes until Study completion at Day 29
  Heart rate data will be collected every 15 minutes over a 4-week period for each participant to identify changes that may be indicative of infection. These data points will be used as input features for a machine learning model aimed at predicting infection risk in children receiving cancer treatment.
Changes in heart rhythm | Baseline (Day 1) and every 15 minutes until Study completion at Day 29
  Detection of irregular heart rhythms that may reflect early signs of infection. These data points will be used as input features for a machine learning model aimed at predicting infection risk in children receiving cancer treatment.
Changes in blood oxygen saturation | Baseline (Day 1) and every 15 minutes until Study completion at Day 29
  Blood oxygen saturation data will be collected every 15 minutes over a 4-week period for each participant to identify changes that may be indicative of infection. These data points will be used as input features for a machine learning model aimed at predicting infection risk in children receiving cancer treatment.
Changes in respiratory rate | Baseline (Day 1) and every 15 minutes until Study completion at Day 29
  Respiratory rate data will be collected every 15 minutes over a 4-week period for each participant to identify changes that may be indicative of infection. These data points will be used as input features for a machine learning model aimed at predicting infection risk in children receiving cancer treatment.
Infection-Related Hospital Admission | Baseline (Day 1), Day 8, Day 15, Day 22, Day 29
  An infection survey will be completed by patients once per week over a 4-week period to identify confirmed episodes of infections requiring admission to hospital. This data will be used to determine when patients are controls (non-infectious) vs cases (infectious), and used as an input feature for a machine learning model.

SECONDARY OUTCOMES:
The acceptability of using (and not using) wearable devices in children receiving cancer therapies | Day 29
  The acceptability of using wearable devices in children receiving cancer therapies as determined at study completion using the Theoretical Framework of Acceptability (TFA).

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Children's Hospital, Parkville, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data set collected for this trial will be available 12 months after publication of the primary outcome.
  The study protocol, analysis plan and consent forms will also be available. The data may be obtained from the Murdoch Children's Research Institute by emailing MCTC@mcri.edu.au.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The de-identified data set collected for this trial will be available 12 months after publication of the primary outcome. The data may be obtained from the Murdoch Children's Research Institute by emailing MCTC@mcri.edu.au.
  Prior to accessing any data, the following would be required: a data access agreement must be signed by all relevant parties, the investigators of the study must see and approve the analysis plan describing how the data will be analyzed. There must also be an agreement around appropriate acknowledgement in any future publications.
Access Criteria: The data may be obtained from the Murdoch Children's Research Institute by emailing MCTC@mcri.edu.au.
URL: https://www.mcri.edu.au/research/core-facilities-services/melbourne-children-trials-centre